Cover letter for NCT03328143 Protocol ID 17.101 Protocol title Feasibility of Aromatherapy in an Awake Craniotomy Environment Date: November 21, 2020

The document listed as Protocol Synopsis reflects the full Study Protocol and Statistical Analysis Plan. As this was a feasibility study, we did not prepare a formal study protocol or statistical analysis plan.

Thank you,

Richard A Rovin, MD

## **Protocol Summary**

| Γ | [ |
|---|---|
| Title | A Feasibility Study of Lavender Aromatherapy in |
| _ | an Awake Craniotomy Environment |
| Principal Investigator | Richard A Rovin, MD |
| Research Question(s) | Is it possible to utilize lavender aromatherapy |
| | during awake craniotomy |
| Study Aims and Hypotheses | H <sub>0</sub> : Aromatherapy is technically feasible during |
| | awake neurosurgical procedures |
| | Aim 1: To determine the percent of patients who |
| | would consent to participate |
| | Aim2: To determine the study completion rate |
| | for the consented patients |
| Primary Endpoint(s) | 1. The number of patients consenting to |
| | participate |
| | 2. The number of patients completing the |
| | study |
| Secondary Endpoint(s) | <ol> <li>Anxiety before and after lavender</li> </ol> |
| | aromatherapy intervention |
| | 2. Pain before and after lavender |
| | aromatherapy intervention |
| | 3. Patient's expectation of lavender |
| | aromatherapy |
| | 4. Patient satisfaction with lavender |
| | aromatherapy |
| Study Design | Open label, single arm |
| Study Population | Inclusion Criteria: an adult patient undergoing |
| | clinically indicated cranial neurosurgical |
| | procedure |
| | <b>Exclusion Criteria:</b> allergy to lavender |
| | (Lavandula angustifolia); aversion to lavender |
| | scent; history of asthma or COPD; pregnancy; |
| | history of contact dermatitis following exposure |
| | to cosmetic fragrances |
| Treatment | Inhalation of lavender from a nasal inhaler, prior |
| | to the start of surgery and every 30 minutes |
| | thereafter, or if requested by the patient |
| Method of Randomization | N/A |
| Sample Size Calculation | N/A |
| Outcome Measures | VAS-A, VAS-P, expectancy questionnaire, POPM |
| _ | tool |
| Statistical Analysis | Demographic characteristics were noted using |
| | appropriate descriptive statistics for all |

| | categorical and continuous variables. As both |
|-------------------|-------------------------------------------------------|
| | VAS-A and VAS-P were assessed multiple times |
| | for the same patients, mean scores of these |
| | measures were compared using the repeated |
| | measures analysis of variance (ANOVA), |
| | including multivariate analysis of variance |
| | (MANOVA) tests in the general linear model. |
| | Expectancy questionnaire responses were |
| | analyzed using a 2-sided, paired t-test. Mean |
| | POPM scores were compared using an |
| | independent t-test. An alpha of 0.05 was used for |
| | all statistical tests, and all analyses were done |
| | using SAS® 9.4 (SAS Institute Inc., Cary, NC). |
| Interim Analysis | N/A |
| Subgroup Analysis | N/A |
| Safety | This trial used the U.S. Department of Health and |
| | Human Services' Common Terminology Criteria |
| | for Adverse Events, Version 4.0 (published May |
| | 28, 2009; revised June 14, 2010) for toxicity and |
| | adverse event reporting. |
| Closure | The results will be submitted to medical meetings and |
| | peer reviewed journals |